CLINICAL TRIAL: NCT04006951
Title: Development of a Monocentric and Prospective Clinical and Biological Database in Rectum Cancer
Brief Title: Development of a Clinical and Biological Database in Rectum Cancer
Acronym: BCBRectum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICM-BCB-2014/02
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Rectal Neoplasms
Keywords: Cancer; Colorectal cancer; Biological Specimen Banks
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological collection (Experimental): For all the patients include in the study :
  * Paraffin tissue samples (if applicable) collected during pre-therapeutic rectal biopsy
  * Blood samples collected at different times : Before any treatment and Before surgery if the patient received pre-operative radiochemotherapy
  In parallel to this biological collection, standardized clinical data will be entered into a database
  Interventions: Other: Biological collection

INTERVENTIONS:
Other: Biological collection — Blood samples are collected at different times :
  * Before any treatment
  * After pre-operative radiochemotherapy and before surgery (if applicable)

SUMMARY:
A Clinical and Biological Database will provide to the scientific community a collection of blood and tissues with clinical data to improve knowledge about cancer and help to develope new cancer treatments. This database is specific to Rectum Cancer.

DETAILED DESCRIPTION:
In France, colorectal cancer is the second major cause of cancer-related death with 17 000 cases per year. Rectal carcinoma represents 40% of colorectal cancers.

Locally advanced rectal carcinoma raises the issue of both the oncological control, local and general, and the therapeutic morbidity. Currently, pre-operative radiochemotherapy associated with radical proctectomy (TME) is the standard treatment. Radiochemotherapy improves the local control but with enhanced postoperative morbidity and poor functional results.

Moreover, some patients have no downstaging (around 1/3) and the metastatic risk remains about 30%.

Then, compliance to adjuvant chemotherapy is generally poor after radical proctectomy.

Tumor response to preoperative treatment is the major prognostic factor which reveals tumor aggressiveness. Nevertheless, at present, there are no predictive markers of tumor response.

Progresses in rectal cancer management are related to sharing biological and clinical resources with scientific community.

A clinical and biological collection will allow to :

* develop research programs on predictive markers to pre-operative radiochemotherapy or prognostics factors to disease recurrence
* optimize diagnostic and follow-up tests
* develop new biomarkers to improve patient's therapeutic management

In this context, the Montpellier Cancer Institute (ICM) decided to initiate a biological collection biomedical research dedicated to the tissular and blood samples of patients with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated at the Montpellier Cancer Institute, whatever the treatment received (systemic cancer treatment or radiotherapy or surgery)
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* Patient not affiliated to Social Protection system
* Patient unable to understand or comply with study instructions or requirements for psychological, family, social or geographical reasons
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-10-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who gave their consent to participate in the study | Until the study completion : 66 months
  The proportion of patients who consent to participate in the study among the screened patients

CONTACTS AND LOCATIONS:
Overall Officials: ROUANET Philippe, MD-PhD, Study Chair — Institut régional du Cancer Montpellier
Locations (1):
- ICM Val d'Aurelle, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haustermans K, Debucquoy A, Lambrecht M. The ESTRO Breur Lecture 2010: toward a tailored patient approach in rectal cancer. Radiother Oncol. 2011 Jul;100(1):15-21. doi: 10.1016/j.radonc.2011.05.024. Epub 2011 May 31. PMID 21632132